CLINICAL TRIAL: NCT02952469
Title: Biodistribution and Reproducibility of Ga-68 PSMA-HBED-CC Positron Emission Tomography in Patients With Biopsy Proven Metastatic Prostate Cancer
Brief Title: Biodistribution/Reproducibility Ga-68 PSMA-HBED-CC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201605762
Record Dates: First submitted 2016-10-28; First posted 2016-11-02 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Prostatic Neoplasms
Keywords: Positron-Emission Tomography; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)PSMA-HBED-CC; Glu-NH-CO-NH-Lys-(Ahx)-((68)Ga(HBED-CC)); (68)Ga-PSMA; 68Ga-PSMA-11
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- (68Ga)PSMA-HBED-CC (Experimental): Intervention: positron emission tomography / computed tomography (PET/CT) scan using a experimental radiotracer for imaging prostate-specific membrane antigen
  Interventions: Drug: (68Ga)PSMA-HBED-CC

INTERVENTIONS:
Drug: (68Ga)PSMA-HBED-CC — Experimental radiotracer for imaging prostate cancer
  Other Names: (68Ga)Glu-urea-Lys(Ahx)-HBED-CC

SUMMARY:
The purpose of this Radioactive Drug Research Committee (RDRC) study is to collect initial data regarding biodistribution, reproducibility, and dosimetry for the radiotracer Ga-68 PSMA-HBED-CC, an agent which may be useful for the early detection of metastatic prostate cancer. Investigators will use a test and re-test design in all patients to determine reproducibility of lesion detection and signal intensity, and will include dynamic imaging in some patients for the purposes of dosimetry. Patients with known metastatic prostate cancer will be recruited and imaged on two occasions within the course of 15 days.

DETAILED DESCRIPTION:
Prostate cancer (PCa) represents the most common noncutaneous cancer and second most common cause of cancer related death among men in the United States and worldwide. Individual PCa tumor behavior is variable. Some tumors show slow indolent growth patterns and may never become clinically significant while others are aggressive and lead to metastases and death. PCa most commonly metastasizes to bone and lymph nodes. Lungs, liver, and adrenal glands are less frequent metastatic sites.

Accurate staging and risk stratification is essential to optimal management. Pelvic lymph node dissection (PLND) which is performed along with radical prostatectomy is the gold standard for detection of occult nodal metastases but is invasive and has associated morbidity. PLND offers an additional therapeutic benefit in some patients, but is also associated with potential complications and can still underestimate the extent of nodal metastases as 40-50% fall outside the traditional dissection zones [6]. Furthermore, fewer patients are presenting with nodal metastases at initial presentation due to stage migration, so more PLNDs need to be performed to benefit one patient. Therefore there is a clear need for noninvasive imaging options to assist with early and accurate detection of nodal metastases.

68Ga PSMA-HBED-CC is a urea-based small molecular inhibitor that targets an enzymatic site on the extracellular domain of the PSMA membrane protein. Based on strong preclinical evidence, a number of clinical studies of 68Ga PSMA-HBED-CC PET/CT have been performed. Afshar-Oromieh et al. showed detection of lesions suspicious for PCa metastases in 84% of a cohort of patients (n=37) being investigated for biochemical relapse, clarification of suspicious findings on other modalities, or evaluation for possible 131I PSMA ligands. In a larger retrospective study (n=319) Afshar-Oromieh et al. showed that 68Ga PSMA-HBED-CC PET/CT detected PCa in 83% of patients with suspected recurrence. In another study Afshar-Oromieh et al compared 68Ga PSMA-HBED-CC PET/CT to 18F fluoromethylcholine (FCH) PET/CT. At least one PCa lesion was detected in 87% of patients with 68Ga PSMA-HBED-CC versus 70% of patients with 18F FCH. Among patients in whom PSA values were <2.82 ng/ml at least one lesion could be detected in 69% of patients with 68Ga PSMA-HBED-CC and 44% patients with 18F FCH. Tumor-to-background ratios were higher for 68Ga PSMA-HBED-CC. In the aforementioned studies by Afshar-Oromieh et al. 49 patients with positive scans were further evaluated by biopsy or surgery and were confirmed as PCa with no false positives. Morigi et al. also showed the superiority of 68Ga PSMA-HBED-CC over 18F FCH in PET/CT. Detection rates 68Ga PSMA-HBED-CCPET/CT in multiple studies are higher than for rates reported in the literature for 11C Choline, 18F Choline, and 11C Acetate [20]. Most importantly the detection rates 68Ga PSMA-HBED-CCPET/CT in patients with low PSA (<0.5 ng/ml) are more favorable.

Thus preclinical and clinical studies show that 68Ga PSMA-HBED-CC PET/CT is a promising radiotracer for the early detection of metastatic or recurrent PCa even with low serum PSA levels.

ELIGIBILITY:
There will be no control group. For the study group the following inclusion and exclusion criteria will be followed.

INCLUSION CRITERIA

* Male
* Aged ≥ 18 years
* Histological diagnosis of adenocarcinoma of the prostate OR have a clinical diagnosis of prostate cancer and on active therapy or have received treatment for prostate cancer.
* Multifocal metastatic disease in either castrate sensitive or castrate resistant patients.
* May or may not be on hormonal therapy, chemotherapy, or radium therapy.
* If on hormonal therapy or chemotherapy, must be on it for at least 3 months.
* No plans to undergo prostate cancer therapy administration (with hormone therapy, chemotherapy, radium therapy, external radiation) between the two study exams.
* At least 2 metastatic soft tissue or bone lesions identified on conventional imaging (CT, MRI or bone scan).
* Karnofsky performance status of ≥ 50 (or ECOG/WHO equivalent)
* Ability to understand and willingness to sign a consent document.

EXCLUSION CRITERIA

* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring hospitalization, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Physical limitation that would limit compliance with the study requirements
* Current enrollment in a therapeutic clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Reproducibility assessment | up to 15 days from first imaging
  A second PET imaging assessment will be performed (test/retest) to confirm

SECONDARY OUTCOMES:
Biodistribution assessment | 60 minutes post-injection
  PET imaging assessment of systemic drug distribution using dynamic data

CONTACTS AND LOCATIONS:
Overall Officials: Janet Pollard, M.D., Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afshar-Oromieh A, Avtzi E, Giesel FL, Holland-Letz T, Linhart HG, Eder M, Eisenhut M, Boxler S, Hadaschik BA, Kratochwil C, Weichert W, Kopka K, Debus J, Haberkorn U. The diagnostic value of PET/CT imaging with the (68)Ga-labelled PSMA ligand HBED-CC in the diagnosis of recurrent prostate cancer. Eur J Nucl Med Mol Imaging. 2015 Feb;42(2):197-209. doi: 10.1007/s00259-014-2949-6. Epub 2014 Nov 20. PMID 25411132
- [Background] Jilg CA, Drendel V, Rischke HC, Beck T, Vach W, Schaal K, Wetterauer U, Schultze-Seemann W, Meyer PT. Diagnostic Accuracy of Ga-68-HBED-CC-PSMA-Ligand-PET/CT before Salvage Lymph Node Dissection for Recurrent Prostate Cancer. Theranostics. 2017 Apr 10;7(6):1770-1780. doi: 10.7150/thno.18421. eCollection 2017. PMID 28529650